CLINICAL TRIAL: NCT03455504
Title: Study Investigating Safety, Tolerability and Effectiveness of Venetoclax Add in Combination With Fludarabine, Cyratabine and Idarubicine in Induction of New Onset Non-M3 Acute Myelid Leukemia
Brief Title: Venetoclax Add in Combination With Fludarabine, Cyratabine and Idarubicine in Induction for Acute Myelid Leukemia
Acronym: V-FIRST
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML1718; 2018-000392-33 (EudraCT Number)
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: Study run-in and phase II
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): FLAI + V400 mg
  Interventions: Drug: Venetoclax
- Cohort 2 (Experimental): FLAI + V600 mg
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Venetoclax add in combination with fludarabine, cyratabine and idarubicine

SUMMARY:
This study will test the effectiveness and safety of Venetoclax in combination with standard induction regimen for patients with acute leukemia and poor prognosis.

DETAILED DESCRIPTION:
Intensive treatment of Acute Leukemia, multidrug based chemotherapy induction, achieves complete remission (CR) rates ranging from 50% to 80%. Nonetheless, the majority (60- 70%) of responding patients will eventually relapse.

Patients with non-low risk leukemia according most diffuse risk scores have a poor prognosis and a short survival. For these patient traditional chemotherapy seems to be ineffective, even with BMT consolidation, probably due to activation of survival pathways in Leukemia cells, so that novel therapeutic interventions should be attempted.

This study will test the effectiveness and safety of Venetoclax, a selective BCL2 inhibitor, in combination with standard induction regimen.

Inhibiting anti-apoptotic pathway of BCL2, the investigators expect to improve success rate of standard chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented/confirmed new onset non-m3 acute myeloid leukemia, according to WHO 2017 will be eligible for this study.
* Hematological illness has to be graded intermediate or high risk according ELN criteria
* Patients ≥ 18 years old and ≤ 65 years old
* ECOG performance status ≤ 2.
* Patients with a life expectancy >12 weeks
* Patients may have AML which has arisen from prior therapies or other antecedent disorder
* Adequate hepatic function
* Adequate pancreatic function
* Adequate renal function assessed by: Serum creatinine within reference laboratory ranges or creatinine clearance (by Cockcroft Gault formula, see Appendix 2) ≥ 50 mL/min for patients in whom, in the Investigator's judgment, serum creatinine level may not adequately reflect renal function.
* All non-hematological adverse events must have resolved to NCI-CTCAE Grade ≤ 2 prior to starting therapy.
* Patients must be considered by Investigator suitable to receive combination chemotherapy.
* Combination chemotherapy has not to be considered toxic without expectation of any benefit for the patient
* For females of childbearing potential, a negative pregnancy test must be documented within 72 hours prior to the first study drug administration.
* All patients must be willing to use effective methods of contraception, during the treatment period and for 100 days after the last dose of Venetoclax. Female patients must be postmenopausal (≥ 1 year of amenorrhea), surgically sterile, or they must agree to use 2 adequate methods of contraception with at least one method with a failure rate of

  ≤ 1% per year (e.g., hormonal implants, combined oral contraceptives, vasectomized partner) and the second preferably a physical barrier method of contraception. Oral or injectable contraceptive agents cannot be the sole method of contraception. Male patients must be surgically sterile or agree to use an acceptable method of contraception.
* Patient must be willing to submit the blood sampling and bone marrow sampling for the PK and PD analyses and exploratory biomarkers.
* Ability to understand and willingness to sign an informed consent form.
* Subject must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* Patients with low risk AML according ELN criteria
* Patients with current clinical evidence of CNS leukemia.
* Patients receiving any other investigational or commercial agents or therapies administered with the intention to treat their malignancy with the exception of Hydroxyurea (HU) or 6-Mercaptopurine (6MP) in patients who need to continue this agent to maintain WBC count ≤10,000/mm3. HU and 6MP must be discontinued at the time of initiation of study medications.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study including but not limited at:
* unstable angina
* Patients who are on anti-microbial agents with therapeutic intent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients achieving complete response (CR) after course 1 or course 2 if course 2 is administered (CR + CRi + CRp) | At 24 months from study entry
  Efficacy in new onset, non ELN Low risk AML (safety run-in, part1, and part2). Effectiveness of Venetoclax added in combination with chemotherapy in obtaining Complete remission in new onset, non ELN Low risk AML (safety run-in, part1, and part2).

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, Study Chair — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) Meldola; Fabio Ciceri, Study Director — Istituto S. Raffaele, Milan
Locations (22):
- Italy (22):
  - Ematologia - ASST Papa Giovanni XXIII, Bergamo
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Spedali Civili - Azienda Ospedaliera U.O. Ematologia, Brescia
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - A.O.U. Careggi - Ematologia, Florence
  - Irccs Aou San Martino - Genova - Uo Clinica Ematologica, Genova
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori IRST, Meldola
  - Fondazione Irccs "Istituto Nazionale Tumori" - Milano - Sc Ematologia, Milan
  - Ospedale Niguarda "Ca Granda" SC Ematologia, Milan
  - U.O. Ematologia e Trapianto di Midollo Ist. Scientifico Ospedale San Raffaele, Milan
  - Asl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagani
  - U.O.C. Ematologia e CTMO Az Ospedaliero Universitaria, Parma
  - Fondazione Ircss Policlinico San Matteo - Pavia - Uo Ematologia, Pavia
  - Dipartimento Oncologico - Ospedale S. Maria delle Croci, Ravenna
  - Università degli Studi "Sapienza" Dip. Biotecnologie Cellulari ed Ematologia, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Ististuto Clinico Humanitas - Rozzano - Uo Oncologia Medica Ed Ematologia, Rozzano
  - Aou "San Giovanni Di Dio E Ruggi D'Aragona" - Salerno - Uoc Ematologia E Trapianti Di Cellule Staminali Emopoietiche, Salerno
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Dipartimento di Oncologia ed Ematologia S.C. -Città della Scienza di Torino San Giovanni Battista, Torino
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marconi G, Piciocchi A, Audisio E, Papayannidis C, Cerrano M, Minotti C, Paoloni F, Guolo F, Bocchia M, Rondoni M, Lico A, Carrabba MG, Della Porta MG, Frigeni M, Giaccone L, Beltrami G, Cattaneo C, Di Chio MC, Serio B, Crea E, Freilone R, Capria S, Curti A, Minetto P, la Sala E, Nanni J, Zannetti BA, Simonetti G, Bochicchio MT, Saglio G, Lemoli RM, Venditti A, Vignetti M, Fazi P, Martinelli G. Safety run-in and part 1 of GIMEMA AML1718: venetoclax combined with FLAI as induction treatment in non-low-risk AML. Blood Adv. 2025 May 27;9(10):2542-2552. doi: 10.1182/bloodadvances.2024014901. PMID 40048742
- See also: GIMEMA Foundation — http://www.gimema.it